CLINICAL TRIAL: NCT05011500
Title: Masks Against Surface-Scanning for Radiation Therapy Immobilisation in Head and Neck Cancer (MASSC Study)
Brief Title: Masks Against Surface-Scanning for Radiation Therapy Immobilisation in Head and Neck Cancer (MASSC)
Acronym: MASSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research Antwerp (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CTOR20051GZA
Record Dates: First submitted 2021-04-29; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Neoplasm
Keywords: Radiotherapy; Radiotherapy, Image-Guided
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Starting with closed mask (Experimental): Patient 1-8, receiving radiotherapy for head and neck cancer in this study. Patients will receive 35 fractions of radiotherapy in total. For the first 5 fractions these patients will receive radiotherapy using a closed mask. For the next 5 fractions these patients will receive radiotherapy using an open mask. For the 5 fractions after that these patients will receive radiotherapy using no mask. This schedule repeats for the rest of their treatment.
  Interventions: Radiation: Radiotherapy with Closed Mask; Radiation: Radiotherapy with Open Mask and Surface Scanning; Radiation: Radiotherapy with No Mask
- Starting with open mask (Experimental): Patient 9-16, receiving radiotherapy for head and neck cancer in this study. Patients will receive 35 fractions of radiotherapy in total. For the first 5 fractions these patients will receive radiotherapy using an open mask. For the next 5 fractions these patients will receive radiotherapy using no mask. For the 5 fractions after that these patients will receive radiotherapy using a closed mask. This schedule repeats for the rest of their treatment.
  Interventions: Radiation: Radiotherapy with Closed Mask; Radiation: Radiotherapy with Open Mask and Surface Scanning; Radiation: Radiotherapy with No Mask
- Starting with no mask (Experimental): Patient 17-24, receiving radiotherapy for head and neck cancer in this study. Patients will receive 35 fractions of radiotherapy in total. For the first 5 fractions these patients will receive radiotherapy using no mask. For the next 5 fractions these patients will receive radiotherapy using a closed mask. For the 5 fractions after that these patients will receive radiotherapy using an open mask. This schedule repeats for the rest of their treatment.
  Interventions: Radiation: Radiotherapy with Closed Mask; Radiation: Radiotherapy with Open Mask and Surface Scanning; Radiation: Radiotherapy with No Mask

INTERVENTIONS:
Radiation: Radiotherapy with Closed Mask — Radiotherapy for head and neck cancer, using a closed mask (full thermoplastic mask) to restrict patient movement.
  Other Names: Full thermoplastic mask
Radiation: Radiotherapy with Open Mask and Surface Scanning — Radiotherapy for head and neck cancer, using an open mask to restrict patient movement. Surface Scanning is used to monitor patient movement/positioning.
Radiation: Radiotherapy with No Mask — Radiotherapy for head and neck cancer, without using a mask to restrict patient movement. Surface Scanning is used to monitor patient movement/positioning.

SUMMARY:
The purpose of this study is to investigate the feasibility of using open masks or no masks in combination with optical surface scanning for radiotherapy in patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Histologically confirmed head and neck cancer.
* Patients treated with radiotherapy (RT) as primary treatment.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0-1 as defined in Appendix 3.
* Each subject must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study.
* Patients must be willing to comply with treatment plan and other study procedures

Exclusion Criteria:

* Patients with significantly altered mental status or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study.
* Patients who cannot stay still during fraction because of a disorder (e.g. Parkinson's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Positional Deviation | Positional Deviation will be assessed from start of treatment period to end of treatment period (up to 7 weeks).
  Patient positioning and movement during treatment will be assessed using cone-beam computed tomopgraphy (CBCT). The position of the patient and target volumes measured by CBCT will be compared to computed tomography (CT) scans made during the initial simulation of treatment. CBCT-scans are made right before administering radiation and after radiation has been administered. Translational and rotational deviations will be measured and expressed in millimeters (for translational deviation) and degrees (for rotational deviation).

SECONDARY OUTCOMES:
Patient Distress | Patient distress will be assessed from start of treatment period to end of treatment period (up to 7 weeks).
  Patient Distress, measured every week using the Subjective Units of Distress Scale (SUDs), a scale of 0-10 where a higher number indicates a worse outcome.
Duration of Treatment | Duration of treatment will be assessed from start of treatment period to end of treatment period (up to 7 weeks).
  Duration of treatment (in minutes), registered in radiotherapy software.
Radiotherapy Technician Satisfaction | Radiotherapy technician satisfaction will be assessed from start of treatment period to end of treatment period (up to 7 weeks).
  Personnel satisfaction, questioned weekly using a personnel satisfaction scale from 0 to 10, where a higher number indicates a better outcome.
Radiation Dose | Radiation dose will be assessed from start of treatment period to end of treatment period (up to 7 weeks).
  In vivo dosimetry will be used to asses the accuracy of treatment. Using PerFRACTION™ in vivo dosimetry. Administered radiation doses will be measured for the target volume and expressed in Gray (Gy).

CONTACTS AND LOCATIONS:
Overall Officials: Daan Nevens, PhD, Principal Investigator — Cancer Research Antwerp
Locations (1):
- GZA Ziekenhuizen campus Sint-Augustinus, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Wiant D, Squire S, Liu H, Maurer J, Lane Hayes T, Sintay B. A prospective evaluation of open face masks for head and neck radiation therapy. Pract Radiat Oncol. 2016 Nov-Dec;6(6):e259-e267. doi: 10.1016/j.prro.2016.02.003. Epub 2016 Feb 13. PMID 27025164
- [Background] Li G, Lovelock DM, Mechalakos J, Rao S, Della-Biancia C, Amols H, Lee N. Migration from full-head mask to "open-face" mask for immobilization of patients with head and neck cancer. J Appl Clin Med Phys. 2013 Sep 6;14(5):243-54. doi: 10.1120/jacmp.v14i5.4400. PMID 24036878
- [Background] Zhao B, Maquilan G, Jiang S, Schwartz DL. Minimal mask immobilization with optical surface guidance for head and neck radiotherapy. J Appl Clin Med Phys. 2018 Jan;19(1):17-24. doi: 10.1002/acm2.12211. Epub 2017 Nov 9. PMID 29119677
- [Background] Dekker J, Rozema T, Boing-Messing F, Garcia M, Washington D, de Kruijf W. Whole-brain radiation therapy without a thermoplastic mask. Phys Imaging Radiat Oncol. 2019 Jul 25;11:27-29. doi: 10.1016/j.phro.2019.07.004. eCollection 2019 Jul. PMID 33458273
- [Background] Ali I, Matthiesen C, Algan O, Thompson S, Bogardus C, Herman T, Ahmad S. Quantitative evaluation of increase in surface dose by immobilization thermoplastic masks and superficial dosimetry using Gafchromic EBT film and Monte Carlo calculations. J Xray Sci Technol. 2010;18(3):319-26. doi: 10.3233/XST-2010-0263. PMID 20714089
- [Background] Stieler F, Wenz F, Shi M, Lohr F. A novel surface imaging system for patient positioning and surveillance during radiotherapy. A phantom study and clinical evaluation. Strahlenther Onkol. 2013 Nov;189(11):938-44. doi: 10.1007/s00066-013-0441-z. Epub 2013 Sep 27. PMID 24068172
- [Background] Cervino LI, Pawlicki T, Lawson JD, Jiang SB. Frame-less and mask-less cranial stereotactic radiosurgery: a feasibility study. Phys Med Biol. 2010 Apr 7;55(7):1863-73. doi: 10.1088/0031-9155/55/7/005. Epub 2010 Mar 12. PMID 20224158
- [Background] Bartlett FR, Donovan EM, McNair HA, Corsini LA, Colgan RM, Evans PM, Maynard L, Griffin C, Haviland JS, Yarnold JR, Kirby AM. The UK HeartSpare Study (Stage II): Multicentre Evaluation of a Voluntary Breath-hold Technique in Patients Receiving Breast Radiotherapy. Clin Oncol (R Coll Radiol). 2017 Mar;29(3):e51-e56. doi: 10.1016/j.clon.2016.11.005. Epub 2016 Nov 24. PMID 27890346
- [Background] van Herk M. Errors and margins in radiotherapy. Semin Radiat Oncol. 2004 Jan;14(1):52-64. doi: 10.1053/j.semradonc.2003.10.003. PMID 14752733

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05011500/Prot_SAP_000.pdf